CLINICAL TRIAL: NCT05207787
Title: A Phase 1/2, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Single and Multiple Doses of Oral Administration of HS-10365 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase Ⅰ/Ⅱ Study of the HS-10365 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10365-101
Record Dates: First submitted 2022-01-09; First posted 2022-01-26 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor
Keywords: Advanced solid tumor; RET gene activation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple doses of HS-10365 and 160mg BID (recommended Phase 2 dose) (Experimental): Phase 1 : Multiple doses of HS-10365 for oral administration. Phase 2 : 160 mg BID of HS-10365
  Interventions: Drug: HS-10365

INTERVENTIONS:
Drug: HS-10365 — Single or multiple dose(s) of HS-10365 daily or twice every day. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and/or unequivocal disease progression.

SUMMARY:
HS-10365 is a small molecular, oral potent, selective RET inhibitor. The purpose of this study is to investigate the safety/tolerability、the pharmacokinetic profile and efficacy of HS-10365 in Chinese advanced solid tumor patients.

DETAILED DESCRIPTION:
This is a multicenter, open-label phase 1/2 study in participants with advanced solid tumors, including RET fusion-positive non-small cell lung cancer and other tumors with RET activation. The trial will be conducted in 2 parts: Phase 1 and phase 2. Participants with advanced cancer are eligible if they have progressed on or intolerant to available standard therapies, or no standard or available curative therapy exists. The phase 1 study is a dose-escalation study, which is designed to evaluate the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of single dose and multiple doses of HS-10365 given once every day (QD) or twice every day (BID). A dose of 160 milligrams (mg) twice a day (BID) has been selected as the recommended phase 2 dose (RP2D). Approximately 273 participants with advanced solid tumors harboring a RET gene alteration will be enrolled to one of nine phase 2 cohorts:

Cohort 1: RET fusion non-small cell lung cancer (NSCLC) that has progressed after at least first-line therapy Cohort 2: RET fusion NSCLC not previously treated for metastatic disease Cohort 3: Medullary thyroid carcinoma that has progressed after at least first-line therapy Cohort 4: RET mutation-positive MTC not previously treated for metastatic disease Cohort 5: RET fusion Radioiodine-refractory thyroid cancer Cohort 6: Advanced solid tumors with RET gene fusion except for cohort 1 to 5 Cohort 7: Advanced solid tumors with RET gene abnormalities and drug resistance or intolerance previously treated with RET inhibitors except for cohort 1 to 6 Cohort 8: Advanced solid tumors with RET gene abnormality except for cohort 1 to 7 Cohort 9: NSCLC with RET gene abnormality except for cohort 1 to 2

ELIGIBILITY:
For phase 1:

1. Men or women aged more than or equal to (≥) 18 years.
2. Locally advanced or metastatic cancer patients confirmed by histology or cytology for who that standard treatment is invalid, unavailable or intolerable
3. Enrollment will be restricted to participants with evidence of a RET gene alteration in tumor as determined by local or central testing. And tumor tissue samples should be provided before the first administration for retrospective detection of RET gene status; blood samples are also allowed.
4. At least one extra-cranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0~1.
6. Estimated life expectancy greater than (>) 12 weeks.
7. Men or women should be using adequate contraceptive measures throughout the study; Females should not be breastfeeding at the time of screening, during the study and until 6 months after completion of the study
8. Females must have evidence of non-childbearing potential.
9. Signed and dated Informed Consent Form.

For phase 2:

As for phase 1 with the following modifications:

1. For Cohort 1: Participants must have progressed following at least first-line treatment following platinum-based chemotherapy combined with or sequential PD-1/PD-L1 immunotherapy； For Cohort 2: Recurrence after previous surgical treatment must meet the conditions of having completed radical surgery for at least 6 month； For Cohort 4: Stage III patients with MTC who are unfit/intolerant or refuse radical surgical treatment and have symptoms or rapid disease progression； For Cohort 5: Recurrence after previous surgical treatment must meet the requirements of 12 months or more after the completion of radical surgery;
2. For Cohort 1 and Cohort 2: Enrollment will be restricted to participants with evidence of a RET gene alteration in tumor as determined by central testing.

   For Cohort 3~9: Enrollment will be restricted to participants with evidence of a RET gene alteration in tumor as determined by local or central testing.
3. For Cohort 1 ~7: At least one measurable lesion as defined by RECIST 1.1.

Exclusion Criteria:

1. For Cohort 1 and Cohort 2，patient's cancer has a known primary driver alteration other than RET.
2. For Cohort 1~6 and Cohort 8~9，patients previously treated with a selective RET inhibitor.
3. Treatment with any of the following:

   Previous or current treatment with selective RET inhibitors(except for cohort 7). Any cytotoxic chemotherapy, investigational agents and anticancer drugs within 14 days of the first dose of study drug (except for cohort 3 and 7).

   Radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose.

   Major surgery within 4 weeks of the first dose of study drug.
4. Inadequate bone marrow reserve or organ function.
5. Uncontrolled pleural effusion or ascites or pericardial effusion.
6. Known and untreated, or active central nervous system metastases.
7. Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow the study drug that would preclude adequate absorption of HS-10365.
8. History of hypersensitivity to any active or inactive ingredient of HS-10365 or to drugs with a similar chemical structure or class to HS-10365.
9. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
10. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study.
11. History of neuropathy or mental disorders, including epilepsy and dementia
12. Determined by the physician, any coexisting disease might lead to life threatening complications or avoid the patients from accomplishing the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: To determine the maximum tolerated dose (MTD) or maximum administrated dose(MAD) | Up to 28 days.
  MTD was defined as the previous dose level at which 2 out of 3 subjects or 2 out of 6 subjects experienced a dose limiting toxicity (DLT).
Phase 2: Response Rate (ORR) assessed by independent review committee (IRC) | From the date of first occurrence of complete response (CR) or partial response (PR) on 2 consecutive occasions (≥4 weeks), until the date of disease progression or withdrawal from study, whichever came first, up to 24 months.
  anti-tumor efficacy will be assessed by best radiographic response based on response evaluation criteria in solid tumors at baseline (Day -28 to -1). For patients that continue on repeating 28-Day cycles after the primary evaluation period, progression will be assessed after each 6 weeks before 18 weeks of therapy and then each 12 weeks. ORR is defined as the percentage of patients with a CR or PR that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | From baseline until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0.
Observed maximum plasma concentration (Cmax) after single dose of HS-10365 | From pre-dose to 120 hours after single dose on Day 1
  n the study of single-dose, Cmax will be obtained following administration of a single oral dose of HS-10365 on Day 1 to Day 6.
Observed maximum plasma concentration (Cmax ss) after multiple dose of HS-10365 | From pre-dose to 24 hours after the first dose of multiple dosing on Day 1 of the following 21-Day cycles of therapy
  At multiple-dose, Cmax ss will be obtained on Day 1 of dosing in the following 21-Day cycles of therapy.
Time to reach maximum plasma concentration (Tmax) after single dose of HS-10365 | From pre-dose to 120 hours after single dose on Day 1
  In the study of single-dose, Tmax will be obtained following administration of a single oral dose of HS-10365 on Day 1 to Day 6.
Apparent terminal half-life (T1/2) after single dose of HS-10365 | From pre-dose to 120 hours after single dose on Day 1
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) after single dose of HS-10365 | From pre-dose to 120 hours after single dose on Day 1
  Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
ORR of HS-10365 | From the date of first occurrence of CR or PR on 2 consecutive occasions (≥4 weeks), until the date of disease progression or withdrawal from study, whichever came first, up to 24 months]（Only phase 1）
  Anti-tumor efficacy will be assessed by best radiographic response based on response evaluation criteria in solid tumors at baseline (Day -28 to -1). For patients that continue on repeating 28-Day cycles after the primary evaluation period, progression will be assessed after each 6 weeks before 18 weeks of therapy and then each 12 weeks. ORR is defined as the percentage of patients with a CR or PR that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.
Disease control rate of HS-10365 (DCR) | From the first occurrence of confirmed CR or PR or SD until the date of disease progression or withdrawal from study, whichever came first, up to 24 months.
  Objective response was assessed by RECIST 1.1 thereby to evaluate disease control rate. Disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks).
Duration of response of HS-10365 (DoR) | From the date of the first dose to disease progression or death in patients who achieve CR or PR, whichever came first, up to 24 months.
  Duration of response assessed by RECIST 1.1. Duration of response was defined as the time from when the criteria for CR or PR were first met to the occurrence of a objective disease progression (PD) or death.
Progression-free survival of HS-10365 (PFS) | From the date of the first dose until the date of disease progression or death from any cause, whichever came first, up to 24 months.
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of ﬁrst dose until the documentation of objective PD or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.
Overall survival (OS) | The time from initial administration to death from any cause, up to 4 years
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital, Shanghai JiaoTong University
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China